CLINICAL TRIAL: NCT02319369
Title: A Phase 1 Study of Milademetan (DS 3032b), an Oral MDM2 Inhibitor, In Dose Escalation as a Single Agent and In Dose Escalation/Expansion In Combination With 5 Azacitidine In Subjects With Acute Myelogenous Leukemia (AML) or High Risk Myelodysplastic Syndrome (MDS)
Brief Title: Safety, Tolerability and Pharmacokinetics of Milademetan Alone and With 5-Azacitidine (AZA) in Acute Myelogenous Leukemia (AML) or High-Risk Myelodysplastic Syndrome (MDS)
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: This study was terminated based on a business decision by the Sponsor.
Sponsor: Daiichi Sankyo (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: DS3032-A-U102
Record Dates: First submitted 2014-12-15; First posted 2014-12-18 (Estimated); Results first posted 2021-10-11 (Actual); Last update posted 2021-10-11 (Actual); Status verified 2021-09

CONDITIONS: Acute Myelogenous Leukemia; Myelodysplastic Syndrome
Keywords: High Risk Myelodysplastic Syndrome; Relapsed/Refractory; Newly Diagnosed; Unfit for Chemotherapy
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Myelodysplastic Syndromes; Recurrence | interventions — milademetan; Azacitidine

STUDY DESIGN:
Intervention Model Description: Parts 1 and 1A are sequential, then Part 2 is parallel
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Part 1, Milademetan Alone (Experimental): Participants receive milademetan alone with different dose schedules
  Interventions: Drug: Milademetan
- Part 1A, Milademetan with 5-azacytidine (AZA) (Experimental): Participants receive milademetan in combination with 5-azacytidine (AZA), with different dose schedules
  Interventions: Drug: Milademetan; Drug: AZA
- Part 2, Cohort 1 (Experimental): Participants with refractory or relapsed acute myelogenous leukemia (AML) receive the recommended dose for Part 2 of milademetan or milademetan with5-azacytidine (AZA)
  Interventions: Drug: AZA; Drug: Milademetan
- Part 2, Cohort 2 (Experimental): Participants with newly diagnosed acute myelogenous leukemia (AML) unfit for intensive chemotherapy receive the recommended dose for Part 2 of milademetan or milademetan with 5-azacytidine (AZA)
  Interventions: Drug: AZA; Drug: Milademetan
- Part 2, Cohort 3 (Experimental): Participants with high-risk myelodysplastic syndrome (MDS) receive the recommended dose for Part 2 of milademetan or milademetan with 5-azacytidine (AZA)
  Interventions: Drug: AZA; Drug: Milademetan

INTERVENTIONS:
Drug: Milademetan — Milademetan will be administered daily as oral capsules or as a combination of multiple oral capsules containing 5 mg, 20 mg, 80 mg, and/or 200 mg
  Other Names: Oral MDM2 Inhibitor
  Arms: Part 1, Milademetan Alone; Part 1A, Milademetan with 5-azacytidine (AZA)
Drug: AZA — AZA will be administered at 75 mg/m^2 subcutaneously or intravenously
  Other Names: 5-Azacitidine
  Arms: Part 1A, Milademetan with 5-azacytidine (AZA); Part 2, Cohort 1; Part 2, Cohort 2; Part 2, Cohort 3
Drug: Milademetan — Milademetan will be administered daily as oral capsules or as a combination of multiple oral capsules containing 5, 20, 80, and/or 200 mg. An alternate combination of 30 mg, 80 mg, and/or 100 mg milademetan may be utilized.
  Other Names: Oral MDM2 Inhibitor
  Arms: Part 2, Cohort 1; Part 2, Cohort 2; Part 2, Cohort 3

SUMMARY:
This study will take place in parts:

* Dose Escalation (Part 1): Participants receive milademetan alone with different dose schedules
* Dose Escalation (Part 1A): Participants receive milademetan in combination with 5-azacytidine (AZA), with different dose schedules

The recommended dose for Part 2 will be selected.

* Dose Expansion (Part 2): After Part 1A, participants will receive the recommended Part 2 dose schedule. There will be three groups - those with:

  1. refractory or relapsed acute myelogenous leukemia (AML)
  2. newly diagnosed AML unfit for intensive chemotherapy
  3. high-risk myelodysplastic syndrome (MDS)
* End-of-Study Follow-Up: Safety information will be collected until 30 days after the last treatment. This is the end of the study.

The recommended dose for the next study will be selected.

DETAILED DESCRIPTION:
The primary analysis will occur after all participants have either discontinued the study or completed at least 6 months of treatment. After the primary analysis, the main study will be closed. Participants who are still on study at least 6 months after enrollment of the last participant in the study may be eligible to continue receiving study drug in a separate extension phase of the protocol

ELIGIBILITY:
Inclusion Criteria

1. Has a diagnosis of refractory or relapsed (R/R) AML or high-risk MDS:

   * Part 1 and 1A (Dose Escalation)

     * Participants with R/R AML, OR
     * Participants with untreated, high-risk MDS or participants who have received prior MDS treatment regimens.
     * Participants ≥18 years old.
   * Part 2 (Dose Expansion)

     * Cohort 1: R/R AML

       * Participants who have treatment failure to prior AML therapy or have relapsed after prior AML therapy.
       * Participants ≥18 years old.
     * Cohort 2: Newly diagnosed AML

       * Participants with newly diagnosed AML who are ineligible for intensive induction chemotherapy. Participants must have had no prior AML treatment, with the exceptions of therapy for antecedent hematologic malignancies or hydroxyurea.
       * Participants ≥75 years old, OR Participants between 18 and 74 years old (inclusive) with at least one of the specific protocol-defined comorbidities.
     * Cohort 3: High-risk MDS

       * Participants with untreated, high-risk MDS or who received up to 2 prior MDS treatment regimens.
2. Has an Eastern Cooperative Oncology Group (ECOG) performance status 0 to 2.

   * As an exception, participants with newly diagnosed AML between 18 and 74 years old (inclusive) in Part 2 Cohort 2 with ECOG Performance Status of 3 will be eligible.
3. Has protocol-defined adequate renal, hepatic and blood clotting functions.
4. Is able to provide written informed consent (or authorized representative), comply with protocol visits and procedures, and take oral medication, and does not have any active infection or comorbidity that would interfere with therapy.
5. If female, is either postmenopausal (no menstrual period for a minimum of 12 months), surgically sterile, or, if of childbearing potential, has a negative serum pregnancy test upon entry into this study and is willing to use maximally effective birth control during the period of therapy and for 6 months following the last investigational drug dose.

   * If male, is surgically sterile or willing to use a maximally effective double-barrier contraception method upon enrollment, during the course of the study, and for 6 months following the last investigational drug dose.
6. Is fully informed about their illness and the investigational nature of the study protocol (including foreseeable risks and possible side effects).
7. Signs and dates an Institutional Review Board-approved informed consent form (including Health Insurance Portability and Accountability Act authorization, if applicable) before performance of any study-specific procedures or tests.
8. Is able and willing to provide bone marrow biopsies/aspirates as requested by the protocol.
9. Is willing to undergo malignancy genotyping for TP53 mutation, insertion, or deletion at screening.

Exclusion Criteria

1. Has a diagnosis of acute promyelocytic leukemia.
2. Has a malignancy that is known to contain a non-synonymous mutation, insertion, or deletion in the TP53 gene determined previously or at screening.
3. Has presence of central nervous system (CNS) involvement of leukemia or a history of primary CNS leukemia.
4. Has a second concurrent primary malignancy that required active treatment within the previous 2 years, except for localized cancers that have apparently been cured, such as non-melanoma skin cancer, superficial bladder cancer, or carcinoma in situ of the cervix or breast.
5. Has any condition that would preclude adequate absorption of DS-3032b, including refractory nausea and vomiting, malabsorption, biliary shunt, significant bowel resection, and/or graft-versus-host disease (GVHD) affecting the gut.
6. Has an uncontrolled infection requiring IV antibiotics, antivirals, or antifungals, known human immunodeficiency virus infection, or active hepatitis B or C infection.
7. Has a concomitant medical condition that would increase the risk of toxicity.
8. Has unresolved toxicities from previous anticancer therapy, defined as toxicities (other than alopecia) not yet resolved to NCI-CTCAE Grade ≤ 1, or baseline. Subjects with chronic Grade 2 toxicities may be eligible at the discretion of the Investigator and Sponsor (eg, Grade 2 chemotherapy-induced neuropathy).
9. Has received Hematopoietic Stem Cell Transplantation (HSCT) within 60 days of the first dose of study drugs or has clinically significant GVHD or GVHD requiring initiation of systemic treatment or systemic treatment escalation within 21 days prior to Screening and/or >Grade 1 persistent or clinically significant GVHD or other non-hematologic toxicity related to HCT.
10. Is receiving concomitant treatment with a strong inhibitor or inducer of cytochrome P450 3A4/5.
11. Has received any therapies intended to treat malignancy within 7 days (small molecules) or 21 days (anti-body/immune based biologics) of first receipt of study drugs [except for hydroxyurea, which must be discontinued at least 48 hours (Day -2) prior to study treatment].
12. Had major surgery within 4 weeks prior to study drug treatment.
13. Participated in a therapeutic clinical study within a washout time of 2 weeks or 5 half-lives of the drug/biologic (whichever is longer) before starting study drug treatment under this protocol, or current participation in other therapeutic investigational procedures.
14. Has prolongation of corrected QT interval using Fridericia's method (QTcF) at rest, where the mean QTcF interval is > 480 ms based on triplicate electrocardiograms (ECGs).
15. Is pregnant or breastfeeding.
16. Has substance abuse or medical, psychological, or social conditions that, in the opinion of the Investigator, may interfere with the subject's participation in the clinical study or evaluation of the clinical study results.
17. Prior treatment with an MDM2 inhibitor.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2014-11-25 (Actual); Primary Completion 2020-08-21 (Actual); Study Completion 2020-08-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Leader, Study Director — Daiichi Sankyo
Locations (5):
- United States (5):
  - City of Hope National Medical Center, Duarte, California
  - University of California San Francisco Medical Center, San Francisco, California
  - University of Kansas Cancer Center, Fairway, Kansas
  - Roswell Park Comprehensive Cancer Center, Buffalo, New York
  - M D Anderson Cancer Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) and applicable supporting clinical trial documents may be available upon request at https://vivli.org/. In cases where clinical trial data and supporting documents are provided pursuant to our company policies and procedures, Daiichi Sankyo will continue to protect the privacy of our clinical trial participants. Details on data sharing criteria and the procedure for requesting access can be found at this web address: https://vivli.org/ourmember/daiichi-sankyo/
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Studies for which the medicine and indication have received European Union (EU) and United States (US), and/or Japan (JP) marketing approval on or after 01 January 2014 or by the US or EU or JP Health Authorities when regulatory submissions in all regions are not planned and after the primary study results have been accepted for publication.
Access Criteria: Formal request from qualified scientific and medical researchers on IPD and clinical study documents from clinical trials supporting products submitted and licensed in the United States, the European Union and/or Japan from 01 January 2014 and beyond for the purpose of conducting legitimate research. This must be consistent with the principle of safeguarding study participants' privacy and consistent with provision of informed consent.
URL: https://vivli.org/ourmember/daiichi-sankyo/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 74 participants who met all inclusion criteria and no exclusion criteria were enrolled and treated at 5 clinic sites in the United States.
Pre-assignment Details: Dose escalation of milademetan was used to determine the maximum tolerated dose. A starting dose of 60 mg milademetan was based on safety and tolerability data obtained in the solid tumor or lymphoma first-in-human study of milademetan (Study DS3032-A-U101; NCT01877382).
Groups:
- Cohort 1: Milademetan 60 mg: Participants were administered 60 mg milademetan daily as oral capsules on Days 1 to 21 of a 28-day cycle.
- Cohort 2: Milademetan 90 mg: Participants were administered 90 mg milademetan daily as oral capsules on Days 1 to 21 of a 28-day cycle.
- Cohort 3: Milademetan 120 mg: Participants were administered 120 mg milademetan daily as oral capsules on Days 1 to 21 of a 28-day cycle.
- Cohort 4: Milademetan 160 mg: Participants were administered 160 mg milademetan daily as oral capsules on Days 1 to 21 of a 28-day cycle.
- Cohort 5: Milademetan 210 mg: Participants were administered 210 mg milademetan daily as oral capsules on Days 1 to 21 of a 28-day cycle
- Cohort 6b: Milademetan 160 mg: Participants were administered 160 mg milademetan daily as oral capsules on Days 1 to 7 of a 28-day cycle.
- Cohort 7c: Milademetan 160 mg: Participants were administered 160 mg milademetan daily as oral capsules for 3 of 14 days repeated twice in a 28-day cycle.
- Cohort 8d: Milademetan 160 mg: Participants were administered 160 mg milademetan daily as oral capsules on Days 1 to 14 of a 28-day cycle.
- Cohort 9d: Milademetan 220 mg: Participants were administered 220 mg milademetan daily as oral capsules on Days 1 to 14 of a 28-day cycle.
- Cohort 10e: Milademetan 160 mg + Azacitidine 75 mg/m^2: Participants were administered 160 mg milademetan daily as oral capsules on Days 5 to 14 of a 28-day cycle and azacitidine was administered on Days 1 to 7.
- Cohort 11f: Milademetan 160 mg + Azacitidine 75 mg/m^2: Participants were administered 160 mg milademetan daily as oral capsules on Days 8 to 14 of a 28-day cycle and azacitidine was administered on Days 1 to 7.
- Cohort 12e: Milademetan 200 mg + Azacitidine 75 mg/m^2: Participants were administered 200 mg milademetan daily as oral capsules on Days 5 to 14 of a 28-day cycle and azacitidine was administered on Days 1 to 7.
- Cohort 13f: Milademetan 200 mg + Azacitidine 75 mg/m^2: Participants were administered 200 mg milademetan daily as oral capsules on Days 8 to 14 of a 28-day cycle and azacitidine was administered on Days 1 to 7.
Period: Overall Study
Arm/Group | Cohort 1: Milademetan 60 mg | Cohort 2: Milademetan 90 mg | Cohort 3: Milademetan 120 mg | Cohort 4: Milademetan 160 mg | Cohort 5: Milademetan 210 mg | Cohort 6b: Milademetan 160 mg | Cohort 7c: Milademetan 160 mg | Cohort 8d: Milademetan 160 mg | Cohort 9d: Milademetan 220 mg | Cohort 10e: Milademetan 160 mg + Azacitidine 75 mg/m^2 | Cohort 11f: Milademetan 160 mg + Azacitidine 75 mg/m^2 | Cohort 12e: Milademetan 200 mg + Azacitidine 75 mg/m^2 | Cohort 13f: Milademetan 200 mg + Azacitidine 75 mg/m^2
Started | 7 | 6 | 11 | 8 | 5 | 7 | 3 | 6 | 4 | 9 | 3 | 4 | 1
Completed | 7 | 6 | 11 | 8 | 5 | 7 | 3 | 6 | 4 | 9 | 3 | 4 | 1
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Baseline demographics were assessed in the Enrolled Analysis Set.
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1: Milademetan 60 mg | Cohort 2: Milademetan 90 mg | Cohort 3: Milademetan 120 mg | Cohort 4: Milademetan 160 mg | Cohort 5: Milademetan 210 mg | Cohort 6b: Milademetan 160 mg | Cohort 7c: Milademetan 160 mg | Cohort 8d: Milademetan 160 mg | Cohort 9d: Milademetan 220 mg | Cohort 10e: Milademetan 160 mg + Azacitidine 75 mg/m^2 | Cohort 11f: Milademetan 160 mg + Azacitidine 75 mg/m^2 | Cohort 12e: Milademetan 200 mg + Azacitidine 75 mg/m^2 | Cohort 13f: Milademetan 200 mg + Azacitidine 75 mg/m^2 | Total
Number analyzed (Participants) | 7 | 6 | 11 | 8 | 5 | 7 | 3 | 6 | 4 | 9 | 3 | 4 | 1 | 74
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.0 (14.7) | 63.8 (10.6) | 61.8 (15.6) | 70.4 (6.1) | 69.2 (7.2) | 71.3 (6.4) | 66.7 (7.6) | 61.8 (20.1) | 72.0 (8.2) | 60.3 (19.8) | 49.3 (25.4) | 70.8 (7.1) | 60.0 (NA) — Standard deviation cannot be calculated for 1 patient. | 66.6 (12.1)
Age, Customized [Count of Participants; unit: Participants]
  ≤65 years | 4 | 4 | 5 | 2 | 1 | 1 | 1 | 3 | 1 | 5 | 2 | 1 | 1 | 31
  >65 years | 3 | 2 | 6 | 6 | 4 | 6 | 2 | 3 | 3 | 4 | 1 | 3 | 0 | 43
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 2 | 3 | 3 | 1 | 2 | 1 | 1 | 3 | 6 | 1 | 1 | 1 | 29
  Male | 3 | 4 | 8 | 5 | 4 | 5 | 2 | 5 | 1 | 3 | 2 | 3 | 0 | 45
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 5
  White | 6 | 6 | 9 | 6 | 4 | 6 | 1 | 4 | 4 | 8 | 1 | 4 | 1 | 60
  More than one race | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 5
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 7 | 6 | 11 | 8 | 5 | 7 | 3 | 6 | 4 | 9 | 3 | 4 | 1 | 74

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Dose-Limiting Toxicities (DLTs) Following Administration of Milademetan Alone and In Combination With 5-Azacitidine (AZA)
Description: A DLT was defined as any treatment-emergent adverse event not attributable to disease or disease-related processes occurring during the observation period (Cycle 1) in each dose-level cohort and is Grade (Gr) 3 or higher according to NCI CTCAE Version 5.0 (Version 4.03 before 01 Apr 2018), with these exceptions: for elevations in hepatic function enzymes, a DLT is defined as: Gr ≥3 aspartate aminotransferase (AST)/alanine aminotransferase (ALT) levels lasting >3 days; AST/ALT >5 × ULN if accompanied by ≥Gr 2 elevation in bilirubin. Potential DLTs include: Participants who are unable to complete at least 75% of milademetan or AZA in Cycle 1 as a result of non-disease-related Gr ≥2 events; Persistent bone marrow aplasia in the absence of malignant cell infiltration, and failure to recover a peripheral absolute neutrophil count ≥0.5 × 10^9/L and platelets ≥20 × 10^9/L while withholding study drug, resulting in >2-week delay in initiating Cycle 2.
Time Frame: From the date the participant signed the informed consent form up to 5 years of first participant enrolled
Population: Dose-limiting toxicities were reported in the DLT evaluable set for Cohorts 1, 4, 5, and 9d of Part 1 and Cohort 12e of Part 1a.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Milademetan 60 mg | Cohort 4: Milademetan 160 mg | Cohort 5: Milademetan 210 mg | Cohort 9d: Milademetan 220 mg | Cohort 12e: Milademetan 200 mg + Azacitidine 75 mg/m^2
Number analyzed (Participants) | 5 | 8 | 5 | 3 | 4
Participants
  Participants with TEAEs classified as DLTs | 1 | 2 | 3 | 2 | 2
  Nausea | 0 | 0 | 1 | 2 | 0
  Fatigue | 0 | 0 | 1 | 0 | 2
  Cellulitis | 0 | 0 | 1 | 0 | 0
  Diarrhoea | 0 | 1 | 0 | 0 | 0
  Hypokalaemia | 0 | 1 | 0 | 0 | 0
  Renal failure | 0 | 0 | 1 | 0 | 0
  Vomiting | 1 | 0 | 0 | 0 | 0
  Syncope | 0 | 0 | 0 | 0 | 1

2. Primary Outcome: Number of Participants (≥10%) With Treatment-emergent Adverse Events (TEAEs) Following Administration of Milademetan Alone and In Combination With 5-Azacitidine (AZA)
Description: A treatment-emergent adverse event (TEAE) is defined as an adverse event that emerges during the treatment period (up to 30 days after last dose), having been absent at pre-treatment; or reemerges during treatment, having been present at baseline but stopped prior to treatment; or worsens in severity after starting treatment relative to the pre-treatment state, when the adverse event is continuous.
Time Frame: From the date the participant signed the informed consent form up to 30 days after the last dose in the last participant, up to approximately 6 years of first participant enrolled
Population: Safety events were assessed in the Safety Analysis Set.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Milademetan 60 mg | Cohort 2: Milademetan 90 mg | Cohort 3: Milademetan 120 mg | Cohort 4: Milademetan 160 mg | Cohort 5: Milademetan 210 mg | Cohort 6b: Milademetan 160 mg | Cohort 7c: Milademetan 160 mg | Cohort 8d: Milademetan 160 mg | Cohort 9d: Milademetan 220 mg | Cohort 10e: Milademetan 160 mg + Azacitidine 75 mg/m^2 | Cohort 11f: Milademetan 160 mg + Azacitidine 75 mg/m^2 | Cohort 12e: Milademetan 200 mg + Azacitidine 75 mg/m^2 | Cohort 13f: Milademetan 200 mg + Azacitidine 75 mg/m^2
Number analyzed (Participants) | 7 | 6 | 11 | 8 | 5 | 7 | 3 | 6 | 4 | 9 | 3 | 4 | 1
Participants
  Any TEAEs | 7 | 6 | 11 | 8 | 5 | 7 | 3 | 6 | 4 | 9 | 3 | 4 | 1
  Nausea | 5 | 4 | 8 | 6 | 4 | 3 | 2 | 4 | 3 | 5 | 2 | 2 | 1
  Diarrhoea | 2 | 2 | 8 | 5 | 3 | 4 | 2 | 3 | 3 | 1 | 2 | 1 | 0
  Vomiting | 2 | 1 | 4 | 4 | 3 | 2 | 2 | 3 | 3 | 3 | 2 | 0 | 0
  Fatigue | 2 | 1 | 5 | 5 | 3 | 2 | 0 | 1 | 1 | 3 | 2 | 2 | 0
  Thrombocytopenia | 2 | 1 | 4 | 5 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 3 | 0
  Oedema peripheral | 1 | 0 | 4 | 2 | 1 | 3 | 1 | 1 | 1 | 1 | 1 | 1 | 0
  Anaemia | 2 | 3 | 3 | 3 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Decreased appetite | 2 | 0 | 2 | 3 | 3 | 2 | 0 | 1 | 0 | 3 | 2 | 0 | 0
  Hypokalaemia | 0 | 1 | 1 | 4 | 3 | 2 | 0 | 0 | 1 | 1 | 0 | 1 | 0
  Lung infection | 0 | 1 | 2 | 2 | 0 | 2 | 1 | 1 | 2 | 3 | 3 | 0 | 0
  Neutropenia | 1 | 2 | 2 | 3 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0
  Hypomagnesaemia | 0 | 1 | 3 | 1 | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypotension | 2 | 2 | 2 | 1 | 1 | 0 | 0 | 0 | 1 | 3 | 1 | 1 | 0
  Pneumonia | 3 | 1 | 1 | 3 | 0 | 0 | 0 | 1 | 0 | 3 | 1 | 1 | 0
  Dyspnoea | 0 | 1 | 2 | 1 | 3 | 1 | 0 | 0 | 0 | 3 | 3 | 0 | 0
  Sepsis | 2 | 0 | 1 | 1 | 0 | 1 | 1 | 1 | 1 | 2 | 0 | 0 | 0
  Abdominal pain | 2 | 1 | 0 | 0 | 0 | 2 | 0 | 2 | 0 | 3 | 1 | 1 | 0
  Asthenia | 1 | 0 | 1 | 1 | 2 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Dehydration | 1 | 0 | 1 | 1 | 1 | 1 | 0 | 0 | 1 | 2 | 0 | 0 | 0
  Dizziness | 1 | 1 | 0 | 2 | 2 | 0 | 0 | 0 | 0 | 2 | 1 | 1 | 0
  Febrile neutropenia | 1 | 0 | 3 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hyperuricaemia | 2 | 1 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Malaise | 1 | 0 | 1 | 0 | 1 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0
  Cough | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 3 | 0 | 0
  Constipation | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 1 | 1
  Contusion | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 0 | 0
  Myalgia | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 1 | 0 | 0
  Epistaxis | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0
  Headache | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0
  Hypophosphataemia | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0
  Muscular weakness | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0
  Rash maculo-papular | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0
  Rhinorrhoea | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0
  Alanine aminotransferase increased | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
  Athralgia | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
  Death | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
  Depression | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
  Device-related infection | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
  Escherichia infection | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
  Fluid overload | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
  Hemorrhoids | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
  Hyponatraemia | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
  Insomnia | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
  Oropharyngeal pain | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
  Pancytopenia | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
  Pneumonia fungal | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
  Pyrexia | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0

3. Secondary Outcome: Maximum Plasma Concentration (Cmax) Following Administration of Milademetan Alone
Description: Pharmacokinetic parameter maximum plasma concentration (Cmax) of milademetan was assessed at select time points and the geometric means (coefficient of variation %) are presented.
Time Frame: Predose, 1 hour (hr), 2 hr, 3 hr, 6 hr, 8 hr, 10 hr of Cycle 1, Day 1 (Cohorts 1-9d) and Cycle 1, Day 15 (Cohorts 1-5 and 7c) (each cycle is 28 days)
Population: Pharmacokinetics were assessed in the Pharmacokinetic Analysis Set.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Cohort 1: Milademetan 60 mg | Cohort 2: Milademetan 90 mg | Cohort 3: Milademetan 120 mg | Cohort 4: Milademetan 160 mg | Cohort 5: Milademetan 210 mg | Cohort 6b: Milademetan 160 mg | Cohort 7c: Milademetan 160 mg | Cohort 8d: Milademetan 160 mg | Cohort 9d: Milademetan 220 mg
Number analyzed (Participants) | 7 | 6 | 11 | 8 | 5 | 7 | 3 | 6 | 4
ng/mL
  Cycle 1, Day 1 | 386.0 (42.2) | 342.5 (23.4) | 505.9 (56.8) | 622.3 (94.5) | 747.9 (48.1) | 440.0 (74.7) | 758.1 (44.8) | 657.0 (27.2) | 1607.4 (34.4)
  Cycle 1, Day 15 | 498.5 (40.3) | 562.6 (58.6) | 614.3 (55.3) | 753.8 (79.8) | 1329.2 (21.9) | NA (NA) — Maximum plasma concentration (Cmax) was not measured due to insufficient participants' samples. | 669.2 (46.0) | NA (NA) — Maximum plasma concentration (Cmax) was not measured due to insufficient participants' samples. | NA (NA) — Maximum plasma concentration (Cmax) was not measured due to insufficient participants' samples.

4. Secondary Outcome: Maximum Plasma Concentration (Cmax) Following Administration of Milademetan In Combination With 5-Azacitidine (AZA)
Description: Pharmacokinetic parameter maximum plasma concentration (Cmax) was assessed at select time points and the geometric means (coefficient of variation %) are presented.
Time Frame: Predose, 0.5 hour (hr), 1 hr, 2 hr, 3 hr, 6 hr of Cycle 1, Day 1 (AZA); Predose, 0.5 hr, 1 hr, 2 hr, 3 hr, 4 hr, 6-10 hr of Day 5, Day 7 (predose) (Cohorts 10e and 12e), Day 8 (Cohorts 11f and 13f), and Day 14 (Cohorts 10e-13f) (each cycle is 28 days)
Population: Pharmacokinetics were assessed in the Pharmacokinetic Analysis Set.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Cohort 10e: Milademetan 160 mg + Azacitidine 75 mg/m^2 | Cohort 11f: Milademetan 160 mg + Azacitidine 75 mg/m^2 | Cohort 12e: Milademetan 200 mg + Azacitidine 75 mg/m^2 | Cohort 13f: Milademetan 200 mg + Azacitidine 75 mg/m^2
Number analyzed (Participants) | 9 | 3 | 4 | 1
ng/mL
  Cycle 1, Day 1 | 527.0 (61.9) | NA (NA) — Maximum plasma concentration (Cmax) was not measured due to insufficient participants' samples. | 707.0 (37.7) | NA (NA) — Maximum plasma concentration (Cmax) was not measured due to insufficient participants' samples.
  Cycle 1, Day 5 | 704.8 (57.6) | NA (NA) — Maximum plasma concentration (Cmax) was not measured due to insufficient participants' samples. | 1019.6 (72.2) | NA (NA) — Maximum plasma concentration (Cmax) was not measured due to insufficient participants' samples.
  Cycle 1, Day 7 | 702.5 (46.4) | NA (NA) — Maximum plasma concentration (Cmax) was not measured due to insufficient participants' samples. | 769.8 (46.7) | NA (NA) — Maximum plasma concentration (Cmax) was not measured due to insufficient participants' samples.
  Cycle 1, Day 8 | NA (NA) — Maximum plasma concentration (Cmax) was not measured due to insufficient participants' samples. | 327.5 (51.2) | NA (NA) — Maximum plasma concentration (Cmax) was not measured due to insufficient participants' samples. | 266.0 (NA) — CV% could not be measured for 1 participant sample.
  Cycle 1, Day 14 | 1488.6 (55.2) | 1057.9 (20.4) | 1448.2 (57.2) | 1190.0 (NA) — CV% could not be measured for 1 participant sample.

5. Secondary Outcome: Time to Maximum Concentration (Tmax) Following Administration of Milademetan Alone
Description: Pharmacokinetic parameter time to maximum concentration (Tmax) of milademetan was assessed at select time points.
Time Frame: as for outcome 3
Population: Pharmacokinetic parameters were assessed in the Pharmacokinetic Analysis Set.
Measure: Median (Full Range); unit: hours
Arm/Group | Cohort 1: Milademetan 60 mg | Cohort 2: Milademetan 90 mg | Cohort 3: Milademetan 120 mg | Cohort 4: Milademetan 160 mg | Cohort 5: Milademetan 210 mg | Cohort 6b: Milademetan 160 mg | Cohort 7c: Milademetan 160 mg | Cohort 8d: Milademetan 160 mg | Cohort 9d: Milademetan 220 mg
Number analyzed (Participants) | 7 | 6 | 11 | 8 | 5 | 7 | 3 | 6 | 4
hours
  Cycle 1, Day 1 | 3.00 [2.00 to 6.25] | 4.39 [1.98 to 6.08] | 3.00 [2.00 to 6.25] | 4.50 [1.90 to 6.07] | 3.00 [3.00 to 8.07] | 3.00 [2.05 to 10.00] | 3.08 [2.00 to 6.00] | 4.50 [3.00 to 6.00] | 4.56 [3.00 to 6.17]
  Cycle 1, Day 15 | 3.00 [2.00 to 3.28] | 2.99 [2.00 to 6.00] | 3.00 [2.00 to 6.00] | 2.96 [1.08 to 6.00] | 4.50 [2.92 to 6.00] | NA [NA to NA] — Time to maximum concentration (Tmax) was not measured due to insufficient participants' samples. | 3.04 [3.00 to 3.08] | NA [NA to NA] — Time to maximum concentration (Tmax) was not measured due to insufficient participants' samples. | NA [NA to NA] — Time to maximum concentration (Tmax) was not measured due to insufficient participants' samples.

6. Secondary Outcome: Time to Maximum Concentration (Tmax) Following Administration of Milademetan In Combination With 5-Azacitidine (AZA)
Description: Pharmacokinetic parameter time to maximum concentration (Tmax) was assessed at select time points.
Time Frame: as for outcome 4
Population: Pharmacokinetic parameters were assessed in the Pharmacokinetic Analysis Set.
Measure: Median (Full Range); unit: hours
Groups:
- Cohort 10e: Milademetan 160 mg + Azacitidine 75 mg/m^2: Participants were administered 160 mg milademetan daily as a single oral capsule on Days 5 to 14 of a 28-day cycle and azacitidine was administered on Days 1 to 7.
Arm/Group | Cohort 10e: Milademetan 160 mg + Azacitidine 75 mg/m^2 | Cohort 11f: Milademetan 160 mg + Azacitidine 75 mg/m^2 | Cohort 12e: Milademetan 200 mg + Azacitidine 75 mg/m^2 | Cohort 13f: Milademetan 200 mg + Azacitidine 75 mg/m^2
Number analyzed (Participants) | 9 | 3 | 4 | 1
hours
  Cycle 1, Day 1 | 0.77 [0.48 to 2.00] | NA [NA to NA] — Time to maximum concentration (Tmax) was not measured due to insufficient participants' samples. | 0.51 [0.48 to 0.58] | NA [NA to NA] — Time to maximum concentration (Tmax) was not measured due to insufficient participants' samples.
  Cycle 1, Day 5 | 3.02 [2.05 to 6.07] | NA [NA to NA] — Time to maximum concentration (Tmax) was not measured due to insufficient participants' samples. | 4.41 [2.10 to 8.00] | NA [NA to NA] — Time to maximum concentration (Tmax) was not measured due to insufficient participants' samples.
  Cycle 1, Day 7 | 0.56 [0.48 to 0.98] | NA [NA to NA] — Time to maximum concentration (Tmax) was not measured due to insufficient participants' samples. | 0.58 [0.50 to 1.00] | NA [NA to NA] — Time to maximum concentration (Tmax) was not measured due to insufficient participants' samples.
  Cycle 1, Day 8 | NA [NA to NA] — Time to maximum concentration (Tmax) was not measured due to insufficient participants' samples. | 6.33 [6.07 to 8.97] | NA [NA to NA] — Time to maximum concentration (Tmax) was not measured due to insufficient participants' samples. | 3.08 [3.08 to 3.08]
  Cycle 1, Day 14 | 3.00 [2.05 to 10.00] | 6.05 [3.17 to 8.00] | 5.54 [3.08 to 8.00] | 6.15 [6.15 to 6.15]

7. Secondary Outcome: Trough Plasma Concentration (Ctrough) Following Administration of Milademetan Alone
Description: Pharmacokinetic parameter plasma concentration before next dose (Ctrough) of milademetan was assessed at Cycle 1, Day 15 and the geometric means (coefficient of variation %) are presented.
Time Frame: Predose, 1 hour (hr), 2 hr, 3 hr, 6 hr, 8 hr, 10 hr of Cycle 1, Day 15 (Cohorts 1-5 and 7c) (each cycle is 28 days)
Population: Pharmacokinetic parameters were assessed in the Pharmacokinetic Analysis Set.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Cohort 1: Milademetan 60 mg | Cohort 2: Milademetan 90 mg | Cohort 3: Milademetan 120 mg | Cohort 4: Milademetan 160 mg | Cohort 5: Milademetan 210 mg | Cohort 7c: Milademetan 160 mg
Number analyzed (Participants) | 7 | 6 | 11 | 8 | 5 | 3
ng/mL | 197.13 (23.2) | 229.28 (82.0) | 292.60 (59.7) | 184.60 (279.1) | 507.07 (24.0) | NA (NA) — Trough plasma concentration (Ctrough) was not measured due to insufficient participants' samples.

8. Secondary Outcome: Area Under the Plasma Concentration Curve up to 24 Hours (AUC0-24) Following Administration of Milademetan Alone
Description: Pharmacokinetic parameter area under the plasma concentration curve up to 24 hours (AUC0-24) of milademetan was assessed at select time points and the geometric means (coefficient of variation %) are presented.
Time Frame: as for outcome 3
Population: Pharmacokinetic parameters were assessed in the Pharmacokinetic Analysis Set.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Cohort 1: Milademetan 60 mg | Cohort 2: Milademetan 90 mg | Cohort 3: Milademetan 120 mg | Cohort 4: Milademetan 160 mg | Cohort 5: Milademetan 210 mg | Cohort 6b: Milademetan 160 mg | Cohort 7c: Milademetan 160 mg | Cohort 8d: Milademetan 160 mg | Cohort 9d: Milademetan 220 mg
Number analyzed (Participants) | 7 | 6 | 11 | 8 | 5 | 7 | 3 | 6 | 4
ng*h/mL
  Cycle 1, Day 1 | 4646.7 (47.7) | 4478.1 (31.2) | 6585.4 (54.8) | 8315.1 (101.2) | 9794.0 (39.4) | 7222.5 (43.1) | 10165.6 (64.6) | 8973.9 (28.1) | 20893.9 (23.2)
  Cycle 1, Day 15 | 7244.6 (28.9) | 8392.9 (56.5) | 9854.9 (54.6) | 10710.8 (54.2) | 20330.2 (15.9) | NA (NA) — Area under the plasma concentration curve up to 24 hours (AUC0-24) was not measured due to insufficient participants' samples. | 7714.3 (30.5) | NA (NA) — Area under the plasma concentration curve up to 24 hours (AUC0-24) was not measured due to insufficient participants' samples. | NA (NA) — Area under the plasma concentration curve up to 24 hours (AUC0-24) was not measured due to insufficient participants' samples.

9. Secondary Outcome: Area Under the Plasma Concentration Curve up to 24 Hours (AUC0-24) Following Administration of Milademetan In Combination With 5-Azacitidine (AZA)
Description: Pharmacokinetic parameter area under the plasma concentration curve up to 24 hours (AUC0-24) was assessed at select time points and the geometric means (coefficient of variation %) are presented.
Time Frame: Predose, 0.5 hr, 1 hr, 2 hr, 3 hr, 4 hr, 6-10 hr of Cycle 1, Day 5 (Cohorts 10e and 12e) and Predose of Cycle 1, Day 14 (Cohorts 10e, 11f, and 12e) (each cycle is 28 days)
Population: Pharmacokinetic parameters were assessed in the Pharmacokinetic Analysis Set.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Cohort 10e: Milademetan 160 mg + Azacitidine 75 mg/m^2 | Cohort 11f: Milademetan 160 mg + Azacitidine 75 mg/m^2 | Cohort 12e: Milademetan 200 mg + Azacitidine 75 mg/m^2
Number analyzed (Participants) | 9 | 3 | 4
ng*h/mL
  Cycle 1, Day 5 | 8238.7 (43.0) | NA (NA) — Area under the plasma concentration curve up to 24 hours (AUC0-24) was not measured due to insufficient participants' samples. | 21299.3 (16.3)
  Cycle 1, Day 14 | 22563.8 (52.9) | 15755.5 (29.4) | 19967.5 (18.5)

10. Secondary Outcome: Serum Macrophage Inhibitory Cytokine-1 (MIC-1) Fold Change From Baseline Following Administration of Milademetan Alone
Description: Pharmacodynamic biomarker serum macrophage inhibitory cytokine-1 (MIC-1) concentrations of milademetan were assessed for Cohorts 1 though 9d. Fold change is the ratio of post-baseline MIC-1 values with respect to the baseline values and is the measure of change of MIC-1 from baseline.
Time Frame: Day 1 (6 hours postdose) up to Day 21-22 (predose), up to approximately 6 years of first participant enrolled
Population: Pharmacodynamic biomarker, MIC-1, was assessed in the Safety Analysis Set.
Measure: Mean (Standard Deviation); unit: fold change
Arm/Group | Cohort 1: Milademetan 60 mg | Cohort 2: Milademetan 90 mg | Cohort 3: Milademetan 120 mg | Cohort 4: Milademetan 160 mg | Cohort 5: Milademetan 210 mg | Cohort 6b: Milademetan 160 mg | Cohort 7c: Milademetan 160 mg | Cohort 8d: Milademetan 160 mg | Cohort 9d: Milademetan 220 mg
Number analyzed (Participants) | 7 | 6 | 11 | 8 | 5 | 7 | 3 | 6 | 4
fold change
  Day 1 (6 hours postdose): number analyzed (Participants) | 7 | 6 | 11 | 8 | 5 | 7 | 3 | 5 | 4
  Day 1 (6 hours postdose) | 3.14 (1.23) | 2.78 (0.95) | 3.36 (1.38) | 3.00 (0.88) | 4.25 (1.41) | 2.64 (0.91) | 3.36 (1.49) | 2.64 (0.87) | 4.94 (2.22)
  Day 2 (predose): number analyzed (Participants) | 7 | 6 | 11 | 8 | 5 | 6 | 3 | 5 | 4
  Day 2 (predose) | 2.53 (0.83) | 3.31 (1.25) | 3.97 (2.71) | 3.44 (1.63) | 5.06 (2.62) | 2.57 (0.81) | 3.84 (1.74) | 3.68 (2.13) | 8.09 (3.27)
  Day 8 (predose): number analyzed (Participants) | 6 | 6 | 9 | 8 | 5 | 7 | 3 | 5 | 4
  Day 8 (predose) | 4.13 (2.46) | 6.35 (4.61) | 7.41 (7.17) | 5.13 (2.64) | 9.70 (7.96) | 4.93 (3.32) | 1.44 (0.36) | 5.63 (3.99) | 13.68 (10.72)
  Day 15 (predose): number analyzed (Participants) | 6 | 6 | 8 | 8 | 5 | 5 | 2 | 5 | 4
  Day 15 (predose) | 2.88 (0.64) | 5.64 (4.94) | 6.04 (3.49) | 5.54 (3.49) | 9.28 (7.26) | 1.33 (0.98) | 1.13 (0.41) | 5.02 (2.20) | 6.61 (4.64)
  Day 21-22 (predose): number analyzed (Participants) | 5 | 4 | 6 | 6 | 4 | 1 | 1 | 3 | 3
  Day 21-22 (predose) | 3.49 (1.88) | 4.61 (2.66) | 4.57 (3.53) | 6.57 (4.22) | 5.88 (2.75) | 0.48 (NA) — Only 1 participant available for analysis; SD cannot be calculated. | 1.24 (NA) — Only 1 participant available for analysis; SD cannot be calculated. | 0.83 (0.45) | 1.18 (0.60)

11. Secondary Outcome: Serum Macrophage Inhibitory Cytokine-1 (MIC-1) Fold Change From Baseline Following Administration of Milademetan In Combination With 5-Azacitidine (AZA)
Description: Pharmacodynamic biomarker serum macrophage inhibitory cytokine-1 (MIC-1) concentrations were assessed for Cohorts 10e though 13f. Fold change is the ratio of post-baseline MIC-1 values with respect to the baseline values and is the measure of change of MIC-1 from baseline.
Time Frame: Day 5 (predose) up to Day 22 (predose), up to approximately 6 years of first participant enrolled
Population: Pharmacodynamic biomarker, MIC-1, was assessed in the Safety Analysis Set.
Measure: Mean (Standard Deviation); unit: fold change
Arm/Group | Cohort 10e: Milademetan 160 mg + Azacitidine 75 mg/m^2 | Cohort 11f: Milademetan 160 mg + Azacitidine 75 mg/m^2 | Cohort 12e: Milademetan 200 mg + Azacitidine 75 mg/m^2 | Cohort 13f: Milademetan 200 mg + Azacitidine 75 mg/m^2
Number analyzed (Participants) | 9 | 3 | 4 | 1
fold change
  Day 5 (predose): number analyzed (Participants) | 6 | 0 | 4 | 0
  Day 5 (predose) | 1.65 (0.72) |  | 1.39 (0.36) |
  Day 5 (6 hours postdose): number analyzed (Participants) | 5 | 0 | 4 | 0
  Day 5 (6 hours postdose) | 3.12 (2.38) |  | 6.07 (2.99) |
  Day 14 (predose): number analyzed (Participants) | 4 | 3 | 2 | 0
  Day 14 (predose) | 10.82 (8.26) | 4.06 (0.54) | 8.34 (6.14) |
  Day 22 (predose): number analyzed (Participants) | 5 | 2 | 2 | 1
  Day 22 (predose) | 2.05 (2.34) | 1.38 (0.29) | 1.81 (1.20) | 1.83 (NA) — Only 1 participant available for analysis; SD cannot be calculated.

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events (TEAEs) were collected from the date the participant signed the informed consent form up to 30 days after the last dose of study drug, up to approximately 6 years of first participant enrolled.
Description: A TEAE was defined as an adverse event that emerges during the treatment period (from first dose date till 30 days after last dose date), having been absent at pre-treatment; or reemerges during treatment, having been present at baseline but stopped prior to treatment; or worsens in severity after starting treatment relative to the pre-treatment state, when the adverse event is continuous.
Arm/Group | Cohort 1: Milademetan 60 mg | Cohort 2: Milademetan 90 mg | Cohort 3: Milademetan 120 mg | Cohort 4: Milademetan 160 mg | Cohort 5: Milademetan 210 mg | Cohort 6b: Milademetan 160 mg | Cohort 7c: Milademetan 160 mg | Cohort 8d: Milademetan 160 mg | Cohort 9d: Milademetan 220 mg | Cohort 10e: Milademetan 160 mg + Azacitidine 75 mg/m^2 | Cohort 11f: Milademetan 160 mg + Azacitidine 75 mg/m^2 | Cohort 12e: Milademetan 200 mg + Azacitidine 75 mg/m^2 | Cohort 13f: Milademetan 200 mg + Azacitidine 75 mg/m^2
All-Cause Mortality (participants affected / at risk) | 1/7 | 0/6 | 1/11 | 1/8 | 1/5 | 1/7 | 1/3 | 1/6 | 2/4 | 2/9 | 2/3 | 1/4 | 0/1
Serious Adverse Events (participants affected / at risk) | 4/7 | 5/6 | 9/11 | 5/8 | 5/5 | 4/7 | 2/3 | 3/6 | 2/4 | 9/9 | 3/3 | 4/4 | 0/1
Other Adverse Events (participants affected / at risk) | 7/7 | 6/6 | 11/11 | 8/8 | 5/5 | 7/7 | 3/3 | 6/6 | 4/4 | 9/9 | 3/3 | 4/4 | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1: Milademetan 60 mg (N=7) | Cohort 2: Milademetan 90 mg (N=6) | Cohort 3: Milademetan 120 mg (N=11) | Cohort 4: Milademetan 160 mg (N=8) | Cohort 5: Milademetan 210 mg (N=5) | Cohort 6b: Milademetan 160 mg (N=7) | Cohort 7c: Milademetan 160 mg (N=3) | Cohort 8d: Milademetan 160 mg (N=6) | Cohort 9d: Milademetan 220 mg (N=4) | Cohort 10e: Milademetan 160 mg + Azacitidine 75 mg/m^2 (N=9) | Cohort 11f: Milademetan 160 mg + Azacitidine 75 mg/m^2 (N=3) | Cohort 12e: Milademetan 200 mg + Azacitidine 75 mg/m^2 (N=4) | Cohort 13f: Milademetan 200 mg + Azacitidine 75 mg/m^2 (N=1)
Lung infection (Infections and infestations) | 0 | 0 | 2 | 1 | 0 | 2 | 1 | 1 | 2 | 3 | 3 | 0 | 0
Pneumonia (Infections and infestations) | 2 | 1 | 0 | 3 | 0 | 0 | 0 | 1 | 0 | 2 | 1 | 1 | 0
Sepsis (Infections and infestations) | 2 | 0 | 1 | 1 | 0 | 0 | 1 | 1 | 1 | 2 | 0 | 0 | 0
Bacteraemia (Infections and infestations) | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia fungal (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0
Arthritis bacterial (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Arthritis infective (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Clostridium difficile colitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Device related sepsis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Zygomycosis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 2 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bone marrow failure (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Splenic infarction (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Asthenia (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Mucosal inflammation (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Multi-organ failure (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cardiac failure (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pericardial effusion (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hemorrhage intracranial (Nervous system disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Confusional state (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Psychogenic seizure (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Renal failure (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urinary incontinence (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Human rhinovirus test positive (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hypotension (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Bacterial infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Device-related infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Escherichia infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Liver abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Parainfluenzae virus infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Periorbital cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pneumonia bacterial (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Staphylococcal sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Ileus (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Death (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Stasis dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Swelling face (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Failure to thrive (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Fluid overload (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1: Milademetan 60 mg (N=7) | Cohort 2: Milademetan 90 mg (N=6) | Cohort 3: Milademetan 120 mg (N=11) | Cohort 4: Milademetan 160 mg (N=8) | Cohort 5: Milademetan 210 mg (N=5) | Cohort 6b: Milademetan 160 mg (N=7) | Cohort 7c: Milademetan 160 mg (N=3) | Cohort 8d: Milademetan 160 mg (N=6) | Cohort 9d: Milademetan 220 mg (N=4) | Cohort 10e: Milademetan 160 mg + Azacitidine 75 mg/m^2 (N=9) | Cohort 11f: Milademetan 160 mg + Azacitidine 75 mg/m^2 (N=3) | Cohort 12e: Milademetan 200 mg + Azacitidine 75 mg/m^2 (N=4) | Cohort 13f: Milademetan 200 mg + Azacitidine 75 mg/m^2 (N=1)
Nausea (Gastrointestinal disorders) | 5 | 4 | 8 | 6 | 4 | 3 | 2 | 4 | 3 | 5 | 2 | 2 | 1
Diarrhoea (Gastrointestinal disorders) | 2 | 2 | 8 | 5 | 3 | 4 | 2 | 3 | 3 | 1 | 2 | 1 | 0
Vomiting (Gastrointestinal disorders) | 2 | 1 | 4 | 4 | 3 | 2 | 2 | 3 | 3 | 3 | 2 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 2 | 1 | 0 | 0 | 0 | 2 | 0 | 2 | 0 | 3 | 1 | 1 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 2 | 2 | 1 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 2 | 0 | 0 | 0
Hemorrhoidal hemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Oral disorder (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Toothache (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Duodenitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Flatulence (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastrointestinal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hiatus hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oesophagitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Proctalgia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Rectal hemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tongue ulceration (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 2 | 1 | 5 | 5 | 3 | 2 | 0 | 1 | 1 | 3 | 2 | 2 | 0
Oedema peripheral (General disorders) | 1 | 0 | 4 | 2 | 1 | 3 | 1 | 1 | 1 | 1 | 1 | 1 | 0
Asthenia (General disorders) | 1 | 0 | 1 | 1 | 2 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Malaise (General disorders) | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Gait disturbance (General disorders) | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 1 | 0 | 1 | 0 | 1 | 1 | 0 | 1 | 0 | 1 | 1 | 0 | 0
Chills (General disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Mucosal inflammation (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Localised oedema (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Multi-organ failure (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pain (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Thirst (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lung infection (Infections and infestations) | 0 | 1 | 2 | 2 | 0 | 2 | 1 | 1 | 2 | 3 | 3 | 0 | 0
Pneumonia (Infections and infestations) | 3 | 1 | 1 | 3 | 0 | 0 | 0 | 1 | 0 | 3 | 1 | 1 | 0
Sepsis (Infections and infestations) | 2 | 0 | 1 | 1 | 0 | 1 | 1 | 1 | 1 | 2 | 0 | 0 | 0
Bacteraemia (Infections and infestations) | 0 | 0 | 1 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 2 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oral candidiasis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Pneumonia fungal (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0
Arthritis bacterial (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Arthritis infective (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Candida infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Clostridium difficile colitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Clostridium difficile infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Device-related sepsis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Influenzae (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Periorbital cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Rash pustular (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sialoadenitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Vulvitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Zygomycosis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 2 | 0 | 2 | 3 | 3 | 2 | 0 | 1 | 0 | 3 | 2 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 4 | 3 | 2 | 0 | 0 | 1 | 1 | 0 | 1 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 1 | 3 | 1 | 2 | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 1 | 1 | 1 | 1 | 0 | 0 | 1 | 2 | 0 | 0 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 2 | 1 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperphosphataemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Fluid overload (Metabolism and nutrition disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Hypouricaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tumour lysis syndrome (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Failure to thrive (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 1 | 4 | 5 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 3 | 0
Anaemia (Blood and lymphatic system disorders) | 2 | 3 | 3 | 3 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 1 | 2 | 2 | 3 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 3 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 1 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bone marrow failure (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Coagulopathy (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Increased tendency to bruise (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Lymphadenitis (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Splenic infarction (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2 | 1 | 3 | 1 | 0 | 0 | 0 | 3 | 3 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 4 | 3 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 2 | 0 | 0 | 0
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Choking (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 1 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 0 | 0
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 1 | 0 | 2 | 2 | 0 | 0 | 0 | 0 | 2 | 1 | 1 | 0
Dysgeusia (Nervous system disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0
Haemorrhage intracranial (Nervous system disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 2 | 1 | 0 | 0
Presyncope (Nervous system disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Disturbance in attention (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dysarthria (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Encephalopathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Memory impairment (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Weight decreased (Investigations) | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cardiac murmur (Investigations) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Electrocardiogram QT prolonged (Investigations) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Activated partial thromboplastin time prolonged (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Bacterial test positive (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood bilirubin increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood creatinine increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Blood potassium increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Brain natriuretic peptide increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Human rhinovirus test positive (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Protein total increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Vitamin D decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hypotension (Vascular disorders) | 2 | 2 | 2 | 1 | 1 | 0 | 0 | 0 | 1 | 3 | 1 | 1 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Embolism (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pallor (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 1 | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 2 | 1 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Joint effusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 3 | 1 | 0 | 0
Synovial cyst (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Agitation (Psychiatric disorders) | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0
Confusional state (Psychiatric disorders) | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Depression (Psychiatric disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Dysphoria (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Psychogenic seizure (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sleep disorder (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 3 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Renal failure (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haemoglobinuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nocturia (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Proteinuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Renal failure acute (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Urinary incontinence (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urinary retention (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pericardial effusion (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Supraventricular tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Tachycardia (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Angina pectoris (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cardiac failure (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cardiac tamponade (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Coronary artery disease (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 3 | 0
Acute febrile neutrophilic dermatosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Purpura (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 2 | 0 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cerumen impaction (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hearing impaired (Ear and labyrinth disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Eye pain (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Retinal haemorrhage (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Vision blurred (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hepatosplenomegaly (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Drug hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Graft versus host disease in skin (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Faeces discoloured (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Ileus (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Mouth haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Device-related infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Escherichia infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Bacterial infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Enterocolitis infectious (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Liver abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Parainfluenzae virus infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Peritonitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pneumonia bacterial (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Skin infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Staphylococcal sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Death (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Oedema (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Tenderness (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0
Acidosis (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hidradenitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Stasis dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Swelling face (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pancytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Tooth fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Orthostatic hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Bradycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dysuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Menorrhagia (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-03-06): https://cdn.clinicaltrials.gov/large-docs/69/NCT02319369/Prot_SAP_000.pdf